CLINICAL TRIAL: NCT03879083
Title: The Impact of Rugae Reproduction on Complete Dentures Patients' Satisfaction: A Randomized Crossover Clinical Trial
Brief Title: The Impact of Rugae Reproduction on Complete Dentures Patients' Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Motasum Abu-Awwad, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 10/2019/27400
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: Patients will randomly be allocated to either group A/B or B/A. Group A: Patients receiving a reproduction of their palatal rugae Group B: Patients receiving a smooth palatal surface.
  After insertion, all participants will be followed up for a minimum of 1 week to correct any issues with the dentures and eliminate patient complaints.
  All patients will be recalled at 2 month after insertion to answer questions using the VAS and to fill out the Oral Health Impact Profile-20 EDENT (OHIP-EDENT), and receive the other type of palatal contour.
  After the second periodthe same process will be repeated.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not be aware of which group he/she is interviewing at the assessment session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With reproduction of palatal rugae (Experimental): Participants will receive maxillary complete dentures with a reproduction of the patients's own palatal rugae to the palatal surface.
  Interventions: Other: The removal of the palatal rugae from the complete denture surface
- Without reproduction of palatal rugae (smooth surface) (Active Comparator): Participants will receive maxillary complete dentures with smooth palatal surfaces without a reproduction of the patients's own palatal rugae to the palatal surface.
  Interventions: Other: Addition of palatal rugae to the complete denture surface

INTERVENTIONS:
Other: Addition of palatal rugae to the complete denture surface — The addition and reproduction of the patient's own palatal rugae to the complete maxillary denture palatal surface.
  Arms: Without reproduction of palatal rugae (smooth surface)
Other: The removal of the palatal rugae from the complete denture surface — The removal of the palatal rugae from the complete maxillary denture palatal surface to become a smooth surface
  Arms: With reproduction of palatal rugae

SUMMARY:
The palatal rugae, refer to asymmetrical and irregular elevations of the mucosa located in the anterior third of the palate, on each side of the median palatal raphe and behind the incisive papilla. The lack of the rugae area on the polished areas of the dentures has been suggested to impact phonetics in denture patients. Therefore, the aim of this randomized crossover clinical trial was to compare patients' reported satisfaction with their complete dentures and oral health related quality of life, when provided with a denture with a reproduction of their rugae on the anterior palatal area as opposed to a polished palatal surface.

DETAILED DESCRIPTION:
The use of dentures could impact the patients' phonetics which could impact their speech. Phonetics could be affected by multiple factors such as having a proper occlusal vertical dimension, proper occlusal plane, correctly positioned anterior and posterior teeth, and adequate contouring of the palatal surface. The lack of the rugae area on the polished areas of the dentures has been also suggested to impact phonetics in denture patients.

The palatal rugae, refer to asymmetrical and irregular elevations of the mucosa located in the anterior third of the palate, on each side of the median palatal raphe and behind the incisive papilla. In addition to enhancing phonetics, the precise reproduction of the rugae in the complete dentures has been suggested to enhance mastication, deglutition and better taste perception. However, these suggestions were based on empirical evidence.

Many studies have described methods for replicating the patients rague on complete dentures, however there are no clinical study to ascertain or negate the impact of this procedure. Therefore, the aim of this randomized crossover clinical trial was to compare patients' reported satisfaction with their complete dentures and oral health related quality of life, when provided with a denture with a reproduction of their rugae on the anterior palatal area as opposed to a polished palatal surface. The null hypothesis was that there would be no difference in patients' reported satisfaction rate using visual analogue scale (VAS) and Oral Health Impact Profile for Edentulous Patients (OHIP-EDENT) Questionnaire response between the two types of palatal contours after using each type for one month post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking a set of conventional maxillary and mandibular complete dentures at the University of Jordan Hospital, for the first time or as a replacement of their previous dentures.
* Patients aged between 45 and 80 years old.
* Patients had been completely edentulous for at least 3 months
* Patients without severe underlying medical conditions, neuromascular dysfunction, auditory problems, mental conditions, oral pathology, xerostomia, or tied tongue condition.
* Patients who approved and consented to participation.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Patients' reported overall satisfaction with their dentures | 60 days
  Patients overall satisfaction rate using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').

SECONDARY OUTCOMES:
Patients reported oral health related quality of life | 60 days
  Patients reported oral health related quality of life using the Oral Health Impact Profile for Edentulous Patients (OHIP-EDENT) Questionnaire; The OHIP-EDENT index has 20 items and uses a 0-5 scale where 0 is never and 5 is always. The minimum overall score can be 20 and maximum 100.
Patients' reported overall satisfaction with their dentures during speaking. | 60 days
  Patients overall satisfaction rate during speaking using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').
Patients' reported overall satisfaction with their dentures during eating | 60 days
  Patients overall satisfaction rate during eating using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').
Patients' reported overall satisfaction with their dentures during drinking | 60 days
  Patients overall satisfaction rate during drinking using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').
Patients' reported overall satisfaction with their ability to clean their dentures | 60 days
  Patients overall satisfaction rate with their ability to clean their dentures using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').
Patients' reported overall satisfaction with their phonetics | 60 days
  Patients' reported overall satisfaction with their phonetics using visual analogue scale (a measurement instrument represented in a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured (satisfied and unsatisfied). Orientated from the left 'best' to the right 'worst').

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided